CLINICAL TRIAL: NCT02119637
Title: Effects of Transcranial Magnetic Stimulation (TMS) on Somatosensory Perception
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140100; 14-AT-0100
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2017-10-17

CONDITIONS: Healthy Volunteer
Keywords: Emotion; Tactile Discrimination; Transcranial Magnetic Stimulation (TMS); Somatosensory; Somatosensory Cortex
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Study 1 TMS to S1: Cohort of healthy participants received screening, brain MRI, TMS to S1 and vertex, and somatosensory testing, including 2-point discrimination and gentle brushing.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Device: MRI
- Study 2 TMS targeting S2/insula: Cohort of healthy participants received screening, brain MRI before and after TMS, TMS to S2/insula and vertex, and somatosensory testing, including 2-point discrimination and gentle brushing.
  Interventions: Device: Transcranial magnetic stimulation (TMS); Device: MRI

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — 1 Hz rTMS for 20 minutes. TMS sessions were separated by at least 24 hours.
Device: MRI — Anatomical MRI, resting state MRI and functional MRI using gentle brushing and finger movement

SUMMARY:
Background:

- Different parts of the brain are involved in feeling touch. Researchers want to study whether repetitive magnetic stimulation (rTMS) to the sensory cortex affects how sensation feels. rTMS is a repeated magnetic pulse that interferes with brain activity. It affects a small part of the brain beneath the scalp. Researchers want to find out the role of sensory cortex in sensing different types of touch.

Objectives:

- To find out the role of sensory cortex, a brain area, in sensing different types of touch.

Eligibility:

- Healthy adults ages 18 45.

Design:

* Participants will be pre-screened with a telephone interview. Then they will be screened with physical and psychological exams and a urine test.
* In Session 1, participants will have an MRI brain scan and fill out questionnaires.
* For MRI, a magnetic field and radio waves take pictures of the brain. Participants will lie on a table that slides in and out of a metal cylinder. A coil will be placed over their head. They will perform a task during the scan. The scanner makes loud knocking noises. Participants will get earplugs. They will be in the scanner for up to 60 minutes.
* In Sessions 2 and 3, participants will take urine tests. Their perception of touch will be measured. Then rTMS will be used to stimulate their sensory cortex and scalp for about 20 minutes. Their perception of touch will be measured again.
* For rTMS, a wire coil is held on the scalp. A brief electrical current passes through the coil and creates a magnetic pulse that affects activity in the brain.

DETAILED DESCRIPTION:
This study will test how parts of sensory cortex relate to different aspects of touch sensation. Healthy male and female adults (ages 18-45) will be enrolled. We will use low frequency repetitive transcutaneous magnetic stimulation (rTMS) to temporarily reduce activation in parts of the sensory cortex and will examine the effect of this procedure on perception of touch stimuli. After screening, participants will undergo three testing sessions. Session 1 will involve questionnaires and anatomical and functional MRI scans (non-invasive brain imaging) that will be used for localizing the correct regions to stimulate with the rTMS. Sessions 2 and 3 will involve active and control rTMS and testing of gentle (non-painful) touch sensation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. between 18 and 45 years old
  2. right-handed.
  3. Fluent in English.
  4. able to provide written informed consent.

EXCLUSION CRITEIRA:

1. Has a dermatological condition such as scars, burns, callouses, or tattoos that might influence cutaneous sensibility on the hands
2. Has had recent or permanent injury of upper limbs or amputation or use of prosthetic arm or leg
3. Used recreational drugs within the past month
4. Is pregnant or breastfeeding.
5. Has a current chronic pain condition or has had chronic pain in the past (painful condition lasting more than six months).
6. Has a major medical condition, such as kidney, liver, cardiovascular, autonomic, pulmonary, or neurological problems (including blindness or deafness) or a chronic systemic disease (e.g. diabetes).
7. Has a medical condition potentially affecting somatosensation (e.g. Raynaud s Disease, peripheral neuropathy, or circulatory disorder).
8. Participant has or had psychiatric disorders such as major depression, major anxiety-related problems, substance or alcohol dependence or abuse, post-traumatic stress syndrome, bipolar disorder, psychosis, or suicide attempts or persistent suicide ideation.
9. Has metal implants or fragments in the body as this would make having an MRI scan unsafe. This includes pacemakers, medication pumps, aneurysm clips, metallic prostheses (such as metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal workers may have.
10. Is uncomfortable in closed spaces (has claustrophobia) so that he/she would feel uncomfortable in the MRI machine, or a condition that prevents him/her from lying flat for up to 1 hour or rotating palm up for 15 minutes while lying flat.
11. Weight of 275 pounds or higher.
12. History of head trauma that was diagnosed as a concussion or was associated with loss of consciousness or was associated with loss of consciousness.
13. Personal history of a seizure or first degree relative with a seizure disorder
14. Participation in brain stimulation within one week of any TMS session in this study
15. Use of neuro-active drugs including opioids, antidepressants, anticonvulsants/antiepileptics, antipsychotics, dopamine agonists, sleep or anxiety medications, stimulants like methylphenidate (Ritalin), antihistamines, certain viral medications, or any other medication affecting the central nervous system
16. History of hearing loss
17. Obtained less than 6 hours of sleep the night before either TMS session (will be asked at each TMS session)
18. Consumed more than 16oz of coffee or an energy drink (anything with 500mg caffeine or more) on the day of the TMS session. (Caffeine > 500mg and sleep deprivation can increase seizure risk (Engel J, 2008).
19. Consumed alcohol on the day of the TMS session or shows signs of alcohol intoxication or alcohol withdrawal syndrome
20. Motor threshold over 82% of Magstim output.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04-17; Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
2-point touch discrimination on hand during active and control rTMS sessions | 2 years
  Primary outcome for Study 1. Touched palm with one or two tips separated by 4 distances. Subject reported if he/she felt one or two touches at each separation distance.

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Bushnell, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baron-Cohen S, Wheelwright S, Skinner R, Martin J, Clubley E. The autism-spectrum quotient (AQ): evidence from Asperger syndrome/high-functioning autism, males and females, scientists and mathematicians. J Autism Dev Disord. 2001 Feb;31(1):5-17. doi: 10.1023/a:1005653411471. PMID 11439754
- [Background] Bolognini N, Rossetti A, Casati C, Mancini F, Vallar G. Neuromodulation of multisensory perception: a tDCS study of the sound-induced flash illusion. Neuropsychologia. 2011 Jan;49(2):231-7. doi: 10.1016/j.neuropsychologia.2010.11.015. Epub 2010 Nov 19. PMID 21094177